CLINICAL TRIAL: NCT06464211
Title: The Effect of Family Counseling Program Applied to University Students With Future Anxiety on Anxiety and Conscious Awareness Levels
Brief Title: The Effect of Family Counseling Program on Anxiety and Conscious Awareness Levels
Acronym: not
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Merve Geylani, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MGeylani
Record Dates: First submitted 2024-05-07; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Anxiety; Awareness; Family Therapy; Cognitive Behavioral Therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study was conducted using an experimental pre-test, post-test, follow-up randomized controlled group experimental research design
Masking Description: no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): There were 6 face-to-face sessions with students for 50- 60 minutes/week, and 2 sessions with internet-based video programs with students' families. Cognitive Behavioral Model-Based Family Counseling Program was conducted. At least one parent was asked to participate in the family sessions. After the implementation of the intervention group was completed, the final tests of the scales used in the research were applied again to both the intervention and the control group. After the data of the study were collected, a focus group interview, one of the interview methods used in qualitative research on the effectiveness and organization of a Cognitive Behavioral Model-Based Family Counseling Program, was conducted for 5 students selected from the initiative group and the effectiveness of the program was evaluated.
  Interventions: Behavioral: Cognitive Behavioral Model-Based Family Counseling Program
- control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Cognitive Behavioral Model-Based Family Counseling Program — A Cognitive Behavioral Model-Based Family Counseling Program is a therapeutic approach that focuses on identifying and changing negative thought patterns and behaviors within the family unit, using principles of cognitive-behavioral therapy to improve communication, resolve conflicts, and enhance overall family functioning.
  Arms: experimental group

SUMMARY:
This study investigates the effect of a Cognitive Behavioral Therapy (CBT)-based Family Counseling Program on the anxiety and mindfulness levels of university students experiencing future anxiety. The research highlights the significance of university education in career development, noting the associated biopsychosocial challenges faced by students. These challenges often manifest as future anxiety-a condition characterized by fear, uncertainty, and stress about future prospects, which can impact students' academic performance, social relationships, and overall mental health. Literature reveals that interventions like CBT, mindfulness practices, and family counseling are effective in managing anxiety and enhancing emotional resilience. The program integrates these approaches to provide dual-layer support, addressing individual thought patterns and family dynamics, thus potentially reducing anxiety and increasing mindfulness among students. This study aims to provide a comprehensive understanding of the program's effectiveness in a controlled setting, contributing to both national and international literature on mental health interventions.

DETAILED DESCRIPTION:
This research was conducted as a pre-test, post-test randomized controlled study to determine the effects of a Cognitive Behavioral Therapy (CBT)-based Family Counseling Program on anxiety and mindfulness levels in university students experiencing future anxiety. The study collected data from 20 students, divided equally between 10 participants in the intervention group and 10 in the control group. Data were gathered using a Personal Characteristics Form, the Future Anxiety Scale for University Students, and the Turkish version of the Mindfulness Awareness Scale for Adolescents and Adults.

The intervention group participated in an online CBT-based Family Counseling Program, which was conducted weekly for 8 weeks, each session lasting between 50-60 minutes. For the first 6 weeks, the sessions included only the students, while the last two weeks also involved family members' participation. No intervention was applied to the control group. Both groups were assessed with the aforementioned scales before the intervention and after its conclusion. This study aims to provide insights into the effectiveness of integrating family dynamics into therapeutic practices for reducing anxiety and enhancing mindfulness among students.

ELIGIBILITY:
Inclusion Criteria:

* The level of future anxiety is above 40 points
* No problems with speech, perception or hearing

  * The person or persons who will be included in the study from family members will be able to participate in the online session at the time required for counseling
  * The student will regularly participate in the interview sessions to be held

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Reduction in Future Anxiety Levels | Baseline (at study start) and at 8 weeks post-intervention.
  This measure assesses the change in future anxiety levels among university students participating in the Cognitive Behavioral Therapy-based Family Counseling Program. The Future Anxiety Scale for University Students will be used to quantify this change. The scale ranges from a minimum score of 19 to a maximum score of 95. Higher scores indicate an increase in the level of future anxiety.
Improvement in Mindfulness Awareness Levels | Baseline (at study start) and at 8 weeks post-intervention.
  This outcome measures the enhancement in mindfulness awareness levels as determined by the Turkish version of the Mindfulness Awareness Scale for Adolescents and Adults. Changes from baseline to post-intervention will be assessed to determine the effectiveness of the intervention. The scale ranges from a minimum score of 18 to a maximum score of 90. Higher scores indicate an increase in the level of mindfulness awareness

CONTACTS AND LOCATIONS:
Overall Officials: merve geylani, MSc, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- IstanbulUC, Şişli, Istanbul, Turkey (Türkiye)